CLINICAL TRIAL: NCT01940198
Title: Long-term Atazanavir Experience in a High HIV Caseload Primary Care Practice in Sydney, Australia
Acronym: REfLecT
Status: Completed | Type: Observational
Sponsor: Holdsworth House Medical Practice (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Dr. Mark Bloch, Principal Investigator, Holdsworth House Medical Practice
Other Study IDs: AI424-417 ST
Record Dates: First submitted 2010-06-01; First posted 2013-09-12 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: HIV
Keywords: Atazanavir; long-term; primary care setting; sydney

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study will aim to determine long-term atazanavir experience in a high HIV caseload primary care practice in Sydney, Australia.

DETAILED DESCRIPTION:
This observational study will aim to determine long term atazanavir experience in HIV-1 infected patients in a primary care setting.

3. OBJECTIVES OF THE STUDY i. Primary objective Long-term (2 years or greater) atazanavir experience in HIV-1 infected patients in a primary care setting through retrospective data collection.

ii. Secondary objectives

1. To illustrate long term therapeutic efficacy of atazanavir in ART naïve and experienced HIV-1 infected patients.
2. To illustrate long term tolerability to atazanavir in ART naïve and experienced HIV-1 infected patients.
3. To identify ART treatment history in ART naïve and experienced HIV-1 infected patients on ATV.
4. To identify contraindicated therapy in ART naïve and experienced HIV-1 infected patients on ATV.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 positive
2. Have commenced ATV between 2002-2008 (Baseline)
3. Follow-up data (clinical and laboratory) available from baseline

Exclusion Criteria:

1. Patients not commenced ATV between 2002-2008
2. No follow-up data (clinical and laboratory) available from baseline
3. Patient 'lost to follow-up' with < 2 years of follow-up data (Clinical and laboratory)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of HIV-1 positive patients attending Holdsworth House Medical Practice who have commenced ATV as a component of ART will be identified from review of current database.
  Data will be collected retrospectively from patient electronic medical records for HIV-1 positive patients that have commenced ATV from year 2002 - 2008.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Proportion of HIV-1 infected participants with atazanavir experience | 1 year
  Proportion of patients who continue on atazanavir for 2 years or greater from baseline to termination/current.

SECONDARY OUTCOMES:
Proportion of HIV-1 infected participants with atazanavir experience | 1 year
  1. Therapeutic efficacy of atazanavir
Proportion of HIV-1 infected participants with atazanavir experience | 1 year
  Tolerability to atazanavir
Proportion of HIV-1 infected participants with atazanavir experience | 1 year
  ART treatment history
Proportion of HIV-1 infected participants with atazanavir experience | 1 year
  contraindicated therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bloch, Dr., Principal Investigator — Holdsworth House Medical Practice
Locations (1):
- Holdsworth House Medical Practice, Sydney, New South Wales, Australia